CLINICAL TRIAL: NCT05452031
Title: A Dyadic Approach to Improve Sleep and Well-Being Among Persons With Alzheimer's Disease and Their Caregivers
Brief Title: A Dyadic Sleep Health Approach for Persons With Alzheimer's Disease and Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of California, San Diego (Other); VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Yeonsu Song, PhD, RN, FNP, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1R01AG076756-01 (NIH)
Record Dates: First submitted 2022-07-01; First posted 2022-07-11 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Sleep
Keywords: Dementia; Caregivers
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-Person Care2Sleep (Experimental): In-person, manual-based sleep hygiene recommendations and a behavioral sleep intervention including sleep compression therapy
  Interventions: Behavioral: Care2Sleep
- Telehealth Care2Sleep (Active Comparator): Telehealth, manual-based sleep hygiene recommendations and a behavioral sleep intervention including sleep compression therapy
  Interventions: Behavioral: Care2Sleep
- Sleep Education only (Placebo Comparator): In-person, education on sleep, aging, and dementia but without specific or individualized recommendations
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: Care2Sleep — A multicomponent behavioral sleep program, consisting of sleep hygiene, stimulus control, sleep compression, pleasurable activity, daily walking, and light exposure.
  Arms: In-Person Care2Sleep; Telehealth Care2Sleep
Behavioral: Sleep Education — This group will receive information about sleep, aging, and dementia, but without specific or individualized recommendations
  Arms: Sleep Education only

SUMMARY:
This is a randomized controlled trial over 5 years, using Stage II of the NIH-defined stage model for behavioral intervention development. We will evaluate the efficacy of the sleep intervention program (Care2Sleep) on sleep, health status measures, and quality of life (for dyads), and inflammation (for caregivers only). Eligible participants will be randomly assigned to in-person Care2Sleep, telehealth Care2Sleep, or to an in-person education control group. The Care2Sleep programs and the control education program will consist of five sessions. The intervention and control programs will begin after baseline assessment and randomization. Posttreatment assessments will be performed immediately after the last session and at 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria for Patients

* Have a diagnosis of Alzheimer's disease (probable or possible) or other related dementia as documented in an electronic medical record
* Community-dwelling
* >1 sleep problems >3x/week on the Neuropsychiatric Inventory Nighttime Behavior Scale, - - Aged >60 years
* Have no untreated sleep disorders (e.g., sleep apnea, restless legs syndrome)
* Able to ambulate with or without assistive devices (i.e., dyads will be excluded if the care recipient is bedbound)
* Have no severe medical conditions with a life expectancy of less than 6 months
* Have an eligible caregiver

Inclusion Criteria for Caregivers

* Live with an eligible patient
* Aged >18 years
* Is related to the patient as a family member, a significant other, or a friend
* Have regularly assisted patient with >1 of 6 basic activities of daily living (ADLs; i.e., bathing, dressing, toileting, transferring, continence, feeding) or >1 of 8 Instrumental ADL (IADLs; i.e., using the telephone, shopping, food preparation, housekeeping, laundry, transportation, taking medications, managing money) for the past 6 months
* Pittsburgh Sleep Quality Index (PSQI) total score >5
* Montreal Cognitive Assessment (MoCA) ≥23
* Can communicate in English

Exclusion Criteria:

* Patients will be excluded if they are bedbound or have severe medical conditions with a life expectancy of less than 6 months.
* Paid, professional caregivers will also be excluded.
* If the eligibility criteria for either a patient or a caregiver are not met, the dyads will be excluded for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Sleep efficiency-Actigraphy | Change from Baseline Sleep Efficiency at 6 months
  Nighttime sleep efficiency (i.e., mean percent of time in bed spent asleep) will be calculated from 7 days of wrist actigraphy for patients and caregivers. Range from 0 to 100% with a higher percent indicating better objective sleep quality
Pittsburgh Sleep Quality Index score | Change from Baseline Pittsburgh Sleep Quality Index score at 6 months
  Self-reported sleep quality over the past week for patients (reported by caregivers) and caregivers. Range from 0 to 21 with lower scores indicating better subjective sleep quality.

SECONDARY OUTCOMES:
Total score of Revised Memory and Behavior Problem Checklist | Immediately AND 6 months after the last session of the intervention
  Dementia-related problem behaviors among persons with dementia (reported by caregivers). Range from 0 to 96 with higher scores indicating more severe dementia-related behaviors.
Total score of Quality of Life-Alzheimer's Disease Scale | Immediately AND 6 months after the last session of the intervention
  Quality of life among persons with dementia reported by either caregivers or persons with dementia. Range from 4 to 52 with higher scores indicating better quality of life among persons with dementia
Total score of Zarit Burden Interview | Immediately AND 6 months after the last session of the intervention
  Perceived levels of caregiving burden. Range from 0 to 88 with higher scores indicating greater burden among caregivers
Total score of Center for Epidemiological Study of Depression Scale | Immediately AND 6 months after the last session of the intervention
  Perceived frequency of depressive symptoms during the past week. Ranges from 0 to 60 with higher scores indicating greater levels of depressive symptoms among caregivers
Patient-Reported Outcomes Measurement Information System (PROMIS) global health score | Immediately AND 6 months after the last session of the intervention
  Self-reported physical and mental health scores among caregivers. A T-score of 50 represents the mean of the general population. Higher scores indicate better physical and mental health among caregivers
Levels of inflammatory markers | Immediately AND 6 months after the last session of the intervention
  Three key inflammatory markers including C-reactive protein, Tumor necrosis factor-alpha, Interleukin-6 will be collected among caregivers only

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California San Diego, La Jolla, California
  - University of California Los Angeles, Los Angeles, California
  - Veterans Affairs Greater Los Angeles Healthcare System, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
Materials generated under the project will be disseminated in accordance with policies at UCLA and NIH. Data products from this study will be made available without cost to researchers, students, and analysts. The final database (both GAD and LAD) will be managed at the UCLA School of Nursing Research Office Design & Data Core. User registration will be required through the Design & Data Core in order to access or download files.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Research data that documents, supports, and validates research findings and referenced resource from a publication will be made available by on-line publication date unless NIH policy specifies an earlier date.